CLINICAL TRIAL: NCT01381003
Title: Phase I/II Gene Therapy Protocol for X-Linked Chronic Granulomatous Disease
Brief Title: Lentiviral Gene Therapy for X-Linked Chronic Granulomatous Disease (X-CGD)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study is withdrawn before recruting participants, new trial will be multi centre, sponsored by different organisation.
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Biren Patel, Great Ormond Street Hospital for Children NHS Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11-MI-03
Record Dates: First submitted 2011-06-23; First posted 2011-06-27 (Estimated); Last update posted 2012-06-04 (Estimated); Status verified 2012-06

CONDITIONS: Granulomatous Disease, Chronic, X-linked, Variant
Keywords: Chronic Granulomatous Disease; Gene therapy; X-CGD; NADPH-oxidase; gp91-phox
MeSH Terms: conditions — Granulomatous Disease, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pCCLchimGp91s lentiviral vector transduced CD34+ cells (Experimental): pCCLchimGp91s lentiviral vector transduced CD34+ cells will be infused in a volume of 50-100 mls intravenously over 30-45 minutes
  Interventions: Genetic: pCCLchimGp91s lentiviral vector transduced CD34+ cells infusion

INTERVENTIONS:
Genetic: pCCLchimGp91s lentiviral vector transduced CD34+ cells infusion — pCCLchimGp91s lentiviral vector transduced CD34+ cells will be infused in a volume of 50-100 mls intravenously over 30-45 minutes

SUMMARY:
Chronic Granulomatous Disease (CGD) is a rare inherited disorder in which patients suffer from severe infection and inflammation. The first indication of disease usually appears in early childhood. The basic defect found to be lie in specialised white blood cells called phagocytic cells, which are responsible for engulfing and destroying germs. In CGD, there is a defect in an enzyme (known as NADPH-oxidase) that is responsible for generating bleach like substances that are important for killing some important germs. In the form of the disease known as X-CGD (which accounts for two thirds of patients), there are defined mistakes in a gene called gp91-phox, which is a key part of the NADPH-oxidase.

In many cases, patients can be protected from infection by constant intake of antibiotics. However, in others potential life-threatening infections break through. In some cases patients also develop serious inflammation requiring high doses of drugs such as steroids. CGD can be cured by bone marrow transplant, but the best results are available when there is matched donor available. Transplant from unmatched donor have a much worse outcome.

Gene therapy of CGD can be performed by introducing a normal copy of human gp91-phox gene into the blood forming stem cells of patients' bone marrow by using a gene carrier (in this study called lentiviral vector). After treatment of the bone marrow cells in a specialised laboratory are given back to the patient and will grow into functional phagocytic cells.

ELIGIBILITY:
Inclusion Criteria:

* History of at least one severe infection requiring hospitalisation despite standard antimicrobial prophylaxis and/or inflammation complications including one of the following: Oesophageal obstruction, gastric outlet obstruction, bladder outlet obstruction or colitis
* Molecular diagnosis confirmed by DNA sequencing and supported by laboratory evidence for absent or significantly reduced biochemical activities of the NADPH-oxidase
* Parental/Guardian and where appropriate Child's signed consent/assent

Exclusion Criteria:

* 10/10 HLA identical (A,B,C,DR,DQ) family or unrelated or cord blood donor unless there is deemed to be an unacceptable risk associated with an allogeneic procedure
* Contraindication for leukapheresis (anaemia Hb <8g/dl, cardiovascular instability, severe coagulopathy) or for administration of conditioning medication

Max Age: 30 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2011-11; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Overall survival following gene therapy | 3 years follow up

SECONDARY OUTCOMES:
Reduction in frequency of infections | evaluated from 1st year after treatment by clinical history, complete physical examination, haematological and microbiological tests
Long term immune reconstitution | 3 years follow up

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Thrasher, Professor, Principal Investigator — Great Ormond Street Hospital for Children NHS Foundation Trust
Locations (1):
- Great Ormond Street Hospital for Children NHS Trust, London, London, United Kingdom